CLINICAL TRIAL: NCT01060449
Title: Stimulus Intensity in Left Ventricular Leads and Response to Cardiac Resynchronization Therapy
Brief Title: Stimulus Intensity in Left Ventricular Leads
Acronym: SILVeR-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Michael S. Lloyd, Principal Investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00016194; Medtronic-639130 (Other: Sponsor)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Congestive Heart Failure
Keywords: cardiac resynchronization therapy; congestive heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LV lead low output (Other): Low output on left ventricular pacing lead.
  Intervention: LV stimulus intensity
  Interventions: Other: LV stimulus intensity
- LV lead high output (Other): High output on left ventricular lead
  Intervention: LV stimulus intensity
  Interventions: Other: LV stimulus intensity

INTERVENTIONS:
Other: LV stimulus intensity — The voltage and pulse duration used for programmed LV pacing
  Arm 1: LV lead low output Arm 2: LV lead high output

SUMMARY:
Cardiac resynchronization therapy (CRT) is a device implanted to improve the function of some people's hearts. CRT involves the placement of 3 wires in the heart through a vein near the front of your left or right shoulder into three pumping chambers of the heart, the most important being the left lower chamber, left ventricle (LV).

DETAILED DESCRIPTION:
The purpose of Cardiac resynchronization therapy (CRT) is to send small amounts of energy (called pacing) through the wires to both the left and right lower chambers of your heart at (or near) the same time. This helps the heart pump in a more coordinated way and send more blood to your body with each beat. How much energy is used for pacing is called the stimulus intensity. Increasing the pacing stimulus intensity of the left ventricular wire can lead to an increase in the volume of heart muscle directly stimulated. This has previously been shown to produce beneficial effects on the heart function, like strength of contraction and increased volume of blood pumped. The purpose of this study is to determine if pacing the wires in the left ventricular chamber of the heart using higher stimulus intensity improves the strength of the heart's contraction.

ELIGIBILITY:
Inclusion Criteria:

* Adults who fulfill approved criteria to receive a cardiac resynchronization device.

Exclusion Criteria:

-Adults who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Ejection Fraction | 6 months

SECONDARY OUTCOMES:
Quality of Life | 6 months
Six minute hall walk | 6 months
End diastolic dimension | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Lloyd, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Bavikati VV, Langberg JJ, Williams BR 3rd, Kella D, Lloyd MS. Stimulus intensity in left ventricular leads and response to cardiac resynchronization therapy. J Am Heart Assoc. 2012 Oct;1(5):e000950. doi: 10.1161/JAHA.112.000950. Epub 2012 Oct 25. PMID 23316285